CLINICAL TRIAL: NCT05790785
Title: Understanding Vascular Complications in Children From Type 1 Diabetes Diagnosis
Brief Title: Vascular Complications in Children From T1D Diagnosis
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Angela Devlin, Professor of Pediatrics, University of British Columbia
Other Study IDs: H21-03109
Record Dates: First submitted 2022-08-04; First posted 2023-03-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes; Cardiovascular Complications; Child; Adolescent
Keywords: Type 1 diabetes; Children; Arterial stiffness; Body composition; Biomarkers; Nutrition; Blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples (20ml) will be collected to evaluate biomarkers of vascular damage. Serum, plasma, and PBMCs will be obtained from the blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with Type 1 diabetes: children recruited within 14 weeks of type 1 diabetes diagnosis and followed for 24 months.

SUMMARY:
Cardiovascular disease is a complication of type 1 diabetes (T1D), a life-long disease, usually diagnosed in childhood. The goal of this project is to determine the timing and factors leading to vascular damage in children from T1D diagnosis.

DETAILED DESCRIPTION:
This is a prospective longitudinal cohort study investigating vascular health in children over the first 2 years of type1 diabetes (T1D) diagnosis living in Metro Vancouver, Canada.

Cardiovascular disease is a major complication of T1D traditionally considered a longterm complication that manifests in adulthood. However, several studies have reported evidence of cardiovascular disease in children who have had T1D for more than 1 year but it is unclear how and when the cardiovascular damage begins. There is also minimal data on cardiovascular complications in children with type 1 diabetes living in Canada.

The goal of this project is to determine the timing and factors leading to vascular damage in children from T1D diagnosis.

We will follow children (aged 8-18 years) from T1D diagnosis over the first 2 years. The primary objective of the study is to assess changes in arterial stiffness (pulse wave velocity; augmentation index), 24-h ambulatory blood pressure (24h-ABPM), and blood biomarkers of vascular damage during the first 2 years of T1D diagnosis.

The secondary objectives of the study are to assess changes in body composition, surrogate markers of adiposity (BMI, waist circumference), and dietary intakes during the first 2 years of T1D diagnosis; and to determine the relationships to measures of arterial stiffness, blood pressure, and blood biomarkers of vascular damage. We will also collect sociodemographic data, estimates of physical activity, and glycated hemoglobin (A1C) as an indicator of glycemic control.

Children with a T1D diagnosis aged 8-18 years will be recruited through the Endocrine and Diabetes Unit at BC Children's Hospital (BCCH). Vascular assessments, blood samples, and data will be collected at diagnosis (within 14 weeks of T1D diagnosis; baseline) and at 6, 12, 18, and 24 months post-diagnosis; there will be a total of 5 visits. Each subject will undergo a clinical assessment, interview/questionnaires, blood collection, and cardiovascular assessment.

Statistical Analysis: . Linear regression models will be used to assess changes in 24-h ABPM mean, daytime and nighttime blood pressure, pulse wave velocity, augmentation index, and biomarkers of vascular damage at diagnosis with values collected during the first 24 months post diagnoses. Models will be adjusted for appropriate covariates. To fully understand the biological differences between males and females, data from boys and girls will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria

1. Between the ages of 8-18 years
2. Within 14 weeks of type 1 diabetes diagnosis
3. Ability and willingness to undergo non-invasive arterial stiffness assessment for 1hr and willingness to wear the 24-h automated blood pressure monitoring (ABPM) device.

Exclusion Criteria

Children will be ineligible to participate in the study if they meet any of the following:

1. Other cardiometabolic or endocrine diseases diagnosis (type 2 diabetes; familial disorders of cholesterol metabolism; lupus)
2. Other genetic syndromes (Down Syndrome; Prader-Willi)
3. Eating disorder diagnosis
4. Transgender children taking hormone blockers or exogenous sex steroids
5. Currently treated with medications known to affect metabolism (e.g. glucocorticoids, antipsychotics).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Transgender children taking hormone blockers or exogenous sex steroids will be excluded because of the potential effect on metabolic health.
Study Population: Children will be recruited within 14 weeks of type 1 diabetes diagnosis through the Endocrine and Diabetes Unit at BC Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in pulse wave velocity during the first 24 months of type 1 diabetes diagnosis | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12, 18 and 24 months post-diagnosis.
  Carotid-femoral pulse wave velocity (PWV) will be measured with a SphygmoCor® XCEL System (AtCor Medical Pty Ltd).
Change in clinic blood pressure during the first 24 months of type 1 diabetes diagnosis | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12, 18 and 24 months post-diagnosis.
  Systolic and diastolic blood pressure measures (average of 3 readings) will be collected using a Dinamap automated monitor (PRO 100-400, GE Medical Systems) and an appropriately sized cuff. Values will be standardized for age, sex, and height using the 2017 American Academy of Pediatrics guidelines.
Change in augmentation index during the first 24 months of type 1 diabetes diagnosis | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Augmentation index will be measured with a SphygmoCor® XCEL System (AtCor Medical Pty Ltd).
Change in 24-h automated blood pressure monitoring (ABPM) during the first 24 months of type 1 diabetes diagnosis | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 12 and 24 months post-diagnosis.
  Children will wear a 24h-ABMP (SpaceLabs) that measures blood pressure every 20 minutes for 24 hours. This will allow for any abnormalities not detected in the clinic to be identified (e.g. masked hypertension). Data will be standardized and categorized according to the 2022 American Academy of Pediatrics guidelines.
Change in biomarkers of vascular health during the first 24 months of type 1 diabetes diagnosis | Baseline (within 14 weeks of type 1 diabetes diagnosis), and at 12 and 24 months post diagnosis.
  Blood biomarkers of vascular health will be assessed in plasma, serum and PBMCs. This includes: a) E-selectin, intracellular adhesion molecule 1 (ICAM), vascular cellular adhesion molecule 1 (VCAM), and von Willebrand factor (vWF) will be quantified as circulating indicators of endothelial damage.
  b) C-reactive protein (CRP), interleukin (IL)-6, IL-8, monocyte chemotactic protein-1 (MCP-1), isoprostane and tumor necrosis factor alpha (TNFα) will be quantified as indicators of inflammation.
  c) Creatinine and total homocysteine will be quantified as indicators of kidney function; d) genome wide DNA methylation patters in PBMCs.

SECONDARY OUTCOMES:
Sociodemographic information | Baseline (within 14 weeks of type 1 diabetes diagnosis). Family history of cardiovascular disease and diabetes and gender will also be assessed at 6, 12, 18, and 24 months.
  Sociodemographic information will be collected including: age, sex, gender, self-reported ethnicity, and family medical history of cardiovascular disease. and diabetes.
Puberty Status | Baseline (within 14 weeks of type 1 diabetes diagnosis), and 12 and 24 months post diagnosis.
  Pubertal development (Tanner stage) will be evaluated by self-reported Tanner staging. The form used for the self-report development stage will be provided to participants according to their sex at birth.
Body weight | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Body weight will be measured measured in children wearing light clothing, pockets emptied, and without shoes using a balance scale. Weight will be recorded to the nearest 0.1 kg.
BMI | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Body mass index (BMI) will be calculated using weight and height measures [weight (kg)/height (m2)] and standardized for sex and age (z-score and percentile) according to WHO growth reference charts.
Physical activity | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Physical activity questionnaire (PAQ) will be administered to quantify relative levels of daily physical activity. There are two versions of the questionnaires: one for elementary school aged children and the second for high school aged children. Participants will be given the questionnaire that corresponds with whether they are in elementary school or high school .
Nutritional assessment | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 12 and 24 months post-diagnosis.
  3x 24-hr dietary recalls will be used to assess dietary intakes. We will conduct 3 dietary recalls for 3 non-consecutive days. The first dietary recall will be will be conducted in person by a member of the research staff during the study visit. The other two diary recalls will be completed over the phone. During the in-person dietary recall, the participants and their parents/caregivers will be shown food models, plates, bowls, cups, and spoons to help them better gauge the amounts of foods and beverages consumed.
Glycated hemoglobin (A1C) | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Blood A1C levels will be measured to assess glycemic control over the past few months. The values for each time point will be obtained from the clinical charts.
  This is routinely done at clinic visits, thus we will obtain this information from medical chart
Body composition | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Body composition will be assessed by Dual-energy X-ray absorptiometry (DEXA) scan (Horizon® Hologic Inc). The percent lean and fat mass and bone density will be calculated from the scans.
Height | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Height will be measured in the children wearing no shoes. Height will be recorded to the nearest 0.1 cm with a stadiometer.
Waist circumference | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Waist circumference will be assessed using a non-elastic flexible tape measure at the level of the umbilicus. The values will be standardized for sex and age (z-score) according to Sharma et al.
Smoking and substance use | Baseline (within 14 weeks of type 1 diabetes diagnosis) and at 6,12,18 and 24 months post-diagnosis.
  Smoking and substance use will be collected as self-reported through direct interview with the subject/family. Collecting this information will allow us to assess the potential impact of smoking habits on vascular health. In addition, tobacco, vaping, e-cigarette, and cannabis use has been described to influence appetite and may affect dietary habits.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Devlin, PhD, Principal Investigator — UBC Pediatrics/BC Children's Hospital Research Institute; Constadina Panagiotopoulos, MD, Principal Investigator — UBC Pediatrics/BC Children's Hospital Research Institute
Locations (1):
- Endocrine and Diabetes Unit, BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the study is completed (Dec 2026).
Access Criteria: Written requests specifying need to access the data should be made to the co-PIs: Dr Angela Devlin and Dr Dina Panagiotopoulos

REFERENCES:
- [Background] Soedamah-Muthu SS, Fuller JH, Mulnier HE, Raleigh VS, Lawrenson RA, Colhoun HM. High risk of cardiovascular disease in patients with type 1 diabetes in the U.K.: a cohort study using the general practice research database. Diabetes Care. 2006 Apr;29(4):798-804. doi: 10.2337/diacare.29.04.06.dc05-1433. PMID 16567818
- [Background] Deckert T, Poulsen JE, Larsen M. Prognosis of diabetics with diabetes onset before the age of thirty-one. I. Survival, causes of death, and complications. Diabetologia. 1978 Jun;14(6):363-70. doi: 10.1007/BF01228130. No abstract available. PMID 669100
- [Background] Secrest AM, Becker DJ, Kelsey SF, Laporte RE, Orchard TJ. Cause-specific mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes. Diabetes. 2010 Dec;59(12):3216-22. doi: 10.2337/db10-0862. Epub 2010 Aug 25. PMID 20739685
- [Background] Krolewski AS, Kosinski EJ, Warram JH, Leland OS, Busick EJ, Asmal AC, Rand LI, Christlieb AR, Bradley RF, Kahn CR. Magnitude and determinants of coronary artery disease in juvenile-onset, insulin-dependent diabetes mellitus. Am J Cardiol. 1987 Apr 1;59(8):750-5. doi: 10.1016/0002-9149(87)91086-1. PMID 3825934
- [Background] Libby P, Nathan DM, Abraham K, Brunzell JD, Fradkin JE, Haffner SM, Hsueh W, Rewers M, Roberts BT, Savage PJ, Skarlatos S, Wassef M, Rabadan-Diehl C; National Heart, Lung, and Blood Institute; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Report of the National Heart, Lung, and Blood Institute-National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Circulation. 2005 Jun 28;111(25):3489-93. doi: 10.1161/CIRCULATIONAHA.104.529651. No abstract available. PMID 15983263
- [Background] Glackin S, Islam N, Henderson AM, Dionne JM, Harris KC, Panagiotopoulos C, Devlin AM. Ambulatory blood pressure and carotid intima media thickness in children with type 1 diabetes. Pediatr Diabetes. 2020 Mar;21(2):358-365. doi: 10.1111/pedi.12960. Epub 2019 Dec 26. PMID 31825119
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Background] Wiltshire EJ, Gent R, Hirte C, Pena A, Thomas DW, Couper JJ. Endothelial dysfunction relates to folate status in children and adolescents with type 1 diabetes. Diabetes. 2002 Jul;51(7):2282-6. doi: 10.2337/diabetes.51.7.2282. PMID 12086961
- [Background] Jarvisalo MJ, Raitakari M, Toikka JO, Putto-Laurila A, Rontu R, Laine S, Lehtimaki T, Ronnemaa T, Viikari J, Raitakari OT. Endothelial dysfunction and increased arterial intima-media thickness in children with type 1 diabetes. Circulation. 2004 Apr 13;109(14):1750-5. doi: 10.1161/01.CIR.0000124725.46165.2C. Epub 2004 Mar 15. PMID 15023875
- [Background] Jarvisalo MJ, Putto-Laurila A, Jartti L, Lehtimaki T, Solakivi T, Ronnemaa T, Raitakari OT. Carotid artery intima-media thickness in children with type 1 diabetes. Diabetes. 2002 Feb;51(2):493-8. doi: 10.2337/diabetes.51.2.493. PMID 11812760
- [Background] Singh TP, Groehn H, Kazmers A. Vascular function and carotid intimal-medial thickness in children with insulin-dependent diabetes mellitus. J Am Coll Cardiol. 2003 Feb 19;41(4):661-5. doi: 10.1016/s0735-1097(02)02894-2. PMID 12598080
- [Background] Krantz JS, Mack WJ, Hodis HN, Liu CR, Liu CH, Kaufman FR. Early onset of subclinical atherosclerosis in young persons with type 1 diabetes. J Pediatr. 2004 Oct;145(4):452-7. doi: 10.1016/j.jpeds.2004.06.042. PMID 15480366
- [Background] Heilman K, Zilmer M, Zilmer K, Lintrop M, Kampus P, Kals J, Tillmann V. Arterial stiffness, carotid artery intima-media thickness and plasma myeloperoxidase level in children with type 1 diabetes. Diabetes Res Clin Pract. 2009 May;84(2):168-73. doi: 10.1016/j.diabres.2009.01.014. Epub 2009 Feb 23. PMID 19237222
- [Background] Ciftel M, Ertug H, Parlak M, Akcurin G, Kardelen F. Investigation of endothelial dysfunction and arterial stiffness in children with type 1 diabetes mellitus and the association with diastolic dysfunction. Diab Vasc Dis Res. 2014 Jan;11(1):19-25. doi: 10.1177/1479164113508564. Epub 2013 Oct 29. PMID 24169808
- [Background] Babar GS, Zidan H, Widlansky ME, Das E, Hoffmann RG, Daoud M, Alemzadeh R. Impaired endothelial function in preadolescent children with type 1 diabetes. Diabetes Care. 2011 Mar;34(3):681-5. doi: 10.2337/dc10-2134. Epub 2011 Feb 2. PMID 21289230
- [Background] Glowinska-Olszewska B, Moniuszko M, Hryniewicz A, Jeznach M, Rusak M, Dabrowska M, Luczynski W, Bodzenta-Lukaszyk A, Bossowski A. Relationship between circulating endothelial progenitor cells and endothelial dysfunction in children with type 1 diabetes: a novel paradigm of early atherosclerosis in high-risk young patients. Eur J Endocrinol. 2013 Jan 17;168(2):153-61. doi: 10.1530/EJE-12-0857. Print 2013 Feb. PMID 23111589
- [Background] Bradley TJ, Slorach C, Mahmud FH, Dunger DB, Deanfield J, Deda L, Elia Y, Har RL, Hui W, Moineddin R, Reich HN, Scholey JW, Mertens L, Sochett E, Cherney DZ. Early changes in cardiovascular structure and function in adolescents with type 1 diabetes. Cardiovasc Diabetol. 2016 Feb 16;15:31. doi: 10.1186/s12933-016-0351-3. PMID 26879273
- [Background] Galler A, Heitmann A, Siekmeyer W, Gelbrich G, Kapellen T, Kratzsch J, Kiess W. Increased arterial stiffness in children and adolescents with type 1 diabetes: no association between arterial stiffness and serum levels of adiponectin. Pediatr Diabetes. 2010 Feb;11(1):38-46. doi: 10.1111/j.1399-5448.2009.00525.x. Epub 2009 May 28. PMID 19496970
- [Background] Duarte SV, de Souza Rajao J, Pinho JF, Dos Santos LM, Alves-Neves CM, Magalhaes GS, Ribeiro-Oliveira A Jr, Rodrigues-Machado MDG. Changes in aortic pulse wave components, pulse pressure amplification, and hemodynamic parameters of children and adolescents with type 1 diabetes. Pediatr Diabetes. 2019 Mar;20(2):202-209. doi: 10.1111/pedi.12782. Epub 2018 Dec 27. PMID 30259609
- [Background] Peppa-Patrikiou M, Scordili M, Antoniou A, Giannaki M, Dracopoulou M, Dacou-Voutetakis C. Carotid atherosclerosis in adolescents and young adults with IDDM. Relation to urinary endothelin, albumin, free cortisol, and other factors. Diabetes Care. 1998 Jun;21(6):1004-7. doi: 10.2337/diacare.21.6.1004. PMID 9614622
- [Background] Rabago Rodriguez R, Gomez-Diaz RA, Tanus Haj J, Avelar Garnica FJ, Ramirez Soriano E, Nishimura Meguro E, Aguilar-Salinas CA, Wacher NH. Carotid intima-media thickness in pediatric type 1 diabetic patients. Diabetes Care. 2007 Oct;30(10):2599-602. doi: 10.2337/dc07-0922. Epub 2007 Jul 20. PMID 17644614
- [Background] Putarek K, Banfic L, Pasalic M, Krnic N, Spehar Uroic A, Rojnic Putarek N. Arterial stiffness as a measure of cardiovascular risk in obese adolescents and adolescents with diabetes type 1. J Pediatr Endocrinol Metab. 2018 Dec 19;31(12):1315-1323. doi: 10.1515/jpem-2018-0137. PMID 30433871
- [Background] Marshall WA, Tanner JM. Variations in pattern of pubertal changes in girls. Arch Dis Child. 1969 Jun;44(235):291-303. doi: 10.1136/adc.44.235.291. No abstract available. PMID 5785179
- [Background] Flynn JT, Urbina EM, Brady TM, Baker-Smith C, Daniels SR, Hayman LL, Mitsnefes M, Tran A, Zachariah JP; Atherosclerosis, Hypertension, and Obesity in the Young Committee of the American Heart Association Council on Lifelong Congenital Heart Disease and Heart Health in the Young; Council on Cardiovascular Radiology and Intervention; Council on Epidemiology and Prevention; Council on Hypertension; and Council on Lifestyle and Cardiometabolic Health. Ambulatory Blood Pressure Monitoring in Children and Adolescents: 2022 Update: A Scientific Statement From the American Heart Association. Hypertension. 2022 Jul;79(7):e114-e124. doi: 10.1161/HYP.0000000000000215. Epub 2022 May 23. PMID 35603599
- [Background] de Onis M, Onyango AW, Borghi E, Siyam A, Nishida C, Siekmann J. Development of a WHO growth reference for school-aged children and adolescents. Bull World Health Organ. 2007 Sep;85(9):660-7. doi: 10.2471/blt.07.043497. PMID 18026621
- [Background] Sharma AK, Metzger DL, Daymont C, Hadjiyannakis S, Rodd CJ. LMS tables for waist-circumference and waist-height ratio Z-scores in children aged 5-19 y in NHANES III: association with cardio-metabolic risks. Pediatr Res. 2015 Dec;78(6):723-9. doi: 10.1038/pr.2015.160. Epub 2015 Sep 2. PMID 26331767
- [Background] Crocker PR, Bailey DA, Faulkner RA, Kowalski KC, McGrath R. Measuring general levels of physical activity: preliminary evidence for the Physical Activity Questionnaire for Older Children. Med Sci Sports Exerc. 1997 Oct;29(10):1344-9. doi: 10.1097/00005768-199710000-00011. PMID 9346166
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, Blowey D, Carroll AE, Daniels SR, de Ferranti SD, Dionne JM, Falkner B, Flinn SK, Gidding SS, Goodwin C, Leu MG, Powers ME, Rea C, Samuels J, Simasek M, Thaker VV, Urbina EM; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017 Sep;140(3):e20171904. doi: 10.1542/peds.2017-1904. Epub 2017 Aug 21. PMID 28827377
- [Background] de Ferranti SD, Steinberger J, Ameduri R, Baker A, Gooding H, Kelly AS, Mietus-Snyder M, Mitsnefes MM, Peterson AL, St-Pierre J, Urbina EM, Zachariah JP, Zaidi AN. Cardiovascular Risk Reduction in High-Risk Pediatric Patients: A Scientific Statement From the American Heart Association. Circulation. 2019 Mar 26;139(13):e603-e634. doi: 10.1161/CIR.0000000000000618. PMID 30798614
- [Background] de Ferranti SD, de Boer IH, Fonseca V, Fox CS, Golden SH, Lavie CJ, Magge SN, Marx N, McGuire DK, Orchard TJ, Zinman B, Eckel RH. Type 1 diabetes mellitus and cardiovascular disease: a scientific statement from the American Heart Association and American Diabetes Association. Circulation. 2014 Sep 23;130(13):1110-30. doi: 10.1161/CIR.0000000000000034. Epub 2014 Aug 11. No abstract available. PMID 25114208
- [Background] Shah AS, Isom S, D'Agostino R, Dolan LM, Dabelea D, Imperatore G, Mottl A, Lustigova E, Pihoker C, Marcovina S, Urbina EM. Longitudinal Changes in Arterial Stiffness and Heart Rate Variability in Youth-Onset Type 1 Versus Type 2 Diabetes: The SEARCH for Diabetes in Youth Study. Diabetes Care. 2022 Jul 7;45(7):1647-1656. doi: 10.2337/dc21-2426. PMID 35667385
- [Derived] Wiedeman AM, Panagiotopoulos C, Devlin AM. Understanding vascular complications in children from type 1 diabetes diagnosis: protocol for a prospective cohort study in Vancouver, Canada. BMJ Open. 2025 Sep 11;15(9):e093842. doi: 10.1136/bmjopen-2024-093842. PMID 40940049